CLINICAL TRIAL: NCT00701220
Title: Statin Induced Augmentation of Circulating Endothelial Progenitor Cells and Myocardial Viability in Patients With Ischemic and Nonischemic Cardiomyopathy
Brief Title: Statin Therapy for Ischemic and Nonischemic Cardiomyopathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Philip Binkley (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Philip Binkley, Professor, Ohio State University
Organization: Ohio State University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005H0118
Record Dates: First submitted 2007-12-26; First posted 2008-06-19 (Estimated); Results first posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-06

CONDITIONS: Cardiovascular Disease; Cardiomyopathy; Heart Disease; Myocardial Disease; Myocardial Ischemia
Keywords: Cardiovascular Disease; Cardiomyopathy; Heart Disease; Myocardial Disease; Myocardial Ischemia
MeSH Terms: conditions — Cardiovascular Diseases; Cardiomyopathies; Heart Diseases; Myocardial Ischemia | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ischemic Cardiomyopathy (Active Comparator): Patients with Ischemic Cardiomyopathy receiving Lipitor (Atorvastatin calcium).
  Interventions: Drug: Atorvastatin Calcium
- Non Ischemic Cardiomyopathy (Active Comparator): NonIschemic Cardiomyopathy receiving Lipitor (Atorvastatin calcium) treatment
  Interventions: Drug: Atorvastatin Calcium
- Healthy Subjects (No Intervention): Healthy subjects with no history of high cholesterol, heart disease, or heart attacks

INTERVENTIONS:
Drug: Atorvastatin Calcium — Atorvastatin Calcium starting at a 10 mg dose and may be increased up to 40 mg dose until cholesterol is lowered to an acceptable range. Blood will drawn every 2 weeks for the first 12 weeks to check the cholesterol level and adjust medication dosage. Cardiac MRI will be performed at the beginning and at the end of the 6 month study to measure the physical changes of the heart.
  Other Names: Lipitor
  Arms: Ischemic Cardiomyopathy; Non Ischemic Cardiomyopathy

SUMMARY:
The purpose of this study is to see if taking a cholesterol lowering drug Lipitor (Atorvastatin Calcium)will increase the number of endothelial progenitor cells (EPC's) circulating in the blood of heart failure patients taking this cholesterol-lowering drug, and if this will also show an improvement in the damaged areas of the patient's hearts as documented by MRI scans.

DETAILED DESCRIPTION:
This study involves the testing of blood for cholesterol levels and flow cytometry tests to count the number of EPC's in your blood. These tests are routinely performed to gain knowledge about a person's health. If any incidental findings are identified as a result of your participation in this research study, you will be notified and referred to your doctor or appropriate health care professional.

You are being asked to provide a blood sample that will be used to determine the usual numbers of EPC's circulating in the blood of healthy people who have no risk factors for heart disease. Your results will be compared with those of patients who have heart failure.

Flow cytometry is a special laboratory test that can count, separate, and detect characteristics of cells in blood. Your blood sample will be analyzed using flow cytometry. Endothelial progenitor cells (EPC's) are immature cells that are necessary for new blood vessel formation. EPC's will be separated by flow cytometry and counted. You will not be given the results of your flow cytometry study.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic Cardiomyopathy (as defined above) with ejection fraction < 35%
* Non-ischemic Cardiomyopathy with ejection fraction < 35%
* NCEP ATPIII indication for therapy with a statin drug
* No statin therapy within previous 6 months of study enrollment
* Prescribed stable doses of standard heart failure therapies including beta blocking agents, angiotensin converting enzyme inhibitors or angiotensin receptor blockers, and diuretic agents as required

Exclusion Criteria:

* Pregnant or lactating
* Myocardial infarction within 6 months preceding study enrollment
* Primary valvular heart disease
* Surgical or catheter based revascularization within the preceding 6 months
* Documented viral or inflammatory myocarditis or cardiomyopathy
* Peripartum cardiomyopathy
* Infiltrative cardiomyopathies
* Chemotherapy associated cardiomyopathy
* Without indication for statin therapy
* Contraindication to statin therapy including hepatic dysfunction, history of rhabdomyolysis or prior intolerance of statin therapy
* Contraindication to magnetic resonance imaging

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Binkley, MD, MPH, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
available through request to the principal investigator; has been presented as an abstract but not a published paper
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Is available now and indefinitely
Access Criteria: Investigators in the field of biomedical research

REFERENCES:
- [Background] Abstract 10678: Increase in the Number of Circulating Primordial Cells is Associated With Improved Left Ventricular Function in Dilated Cardiomyopathy Nkechinyere N Ijioma, Philip F Binkley, and Amanda Lesinski Originally published27 Mar 2018Circulation. 2013;128:A10678

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were eligible for enrollment if they had dilated cardiomyopathy w/ an established ejection fraction < 35% on a nonischemic or ischemic basis. All pts had clinical indication for treatment w/ a statin Rx & did not receive a statin medication prior to enrollment in the study.
Pre-assignment Details: Patients with cardiomyopathy on the basis of valvular heart disease or who had a myocardial infarction within six months prior to study enrollment were excluded from the study.
Groups:
- Ischemic Cardiomyopathy: Patients with Ischemic Cardiomyopathy receiving Lipitor.
- NonIschemic Cardiomyopathy: NonIschemic Cardiomyopathy receiving Lipitor treatment
Period: Overall Study
Arm/Group | Ischemic Cardiomyopathy | NonIschemic Cardiomyopathy
Started | 3 | 6
Completed | 1 | 4
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ischemic Cardiomyopathy | NonIschemic Cardiomyopathy | Total
Number analyzed (Participants) | 1 | 4 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 4 | 5
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.33 (15.29) | 53.66 (9.71) | 52.11 (17.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Endothelial Progenitor Cells
Description: Change in Endothelial Progenitor Cells (EPC) was assessed by extracting white blood cells from blood samples and labeling the white blood cells using the ALDEFLOUR system. Facscan analysis was then performed first isolating lymphocytic and monocytic cell lines, which contain the EPC populations, using forward versus side scatter plots. These cells were then scanned for fluorescence in the ALDEFLUOR frequency range allowing enumeration of progenitor cell lines. The measures of fluorescent cells was compared to numbers of unstained cells having the same back scatter range to correct for any background fluorescence.
Time Frame: Baseline - 6 months
Measure: Mean (Standard Deviation); unit: Percentage of EPCs
Groups:
- NonIschemic Cardiomyopathy: NonIschemic Cardiomyopathy receiving Lipitor (Atorvastatin Calcium) treatment
Arm/Group | Ischemic Cardiomyopathy | NonIschemic Cardiomyopathy
Number analyzed (Participants) | 1 | 4
Percentage of EPCs | -10.01 (0) | 5.19 (0.517)

2. Primary Outcome: Percentage Aldofluor Positive Cells
Description: The primary outcome measure is the percentage of cells of total analyzed that are positive for the Aldofluor assay. This commercially available assay tests cells for the enzyme aldehyde dehydrogenase that is expressed in stem cells and other early life cycle undifferentiated cells. It thus provides a measure of circulating primordial cells or cells that may serve as progenitors of destination mature cells. The percentages are designed from Facscan analysis of prepared blood cells and are quantified by quadrants defined by specific fluorescent bands and cell size distribution. The quantification of cells thus defined in the four quadrants is automatically determined by software resident in the facscan analysis system.
Time Frame: Baseline - 6 months
Measure: Mean (Standard Deviation); unit: Percentage Aldefluor positive cells
Arm/Group | Ischemic Cardiomyopathy | NonIschemic Cardiomyopathy
Number analyzed (Participants) | 1 | 4
Percentage Aldefluor positive cells | 6.37 (0) | 5.7 (0.5)
Statistical Analysis 1: Comparison: Ischemic Cardiomyopathy vs NonIschemic Cardiomyopathy; The data were analyzed using analysis of variance for repeated measures with two groups. The repeated measure was the proportion of circulating blood cells that were positive for aldehyde dehydrogenase using the commercially available Aldofluor assay. The two groups were those with ischemic and non-ischemic cardiomyopathy. This analysis permitted both intergroup and intragroup analysis of the change in aldehyde dehydrogenase positive cells; Test type: Superiority or Other; p < 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: Six months
Description: Adverse events obtained by participant examination and interview
Arm/Group | Ischemic Cardiomyopathy | NonIschemic Cardiomyopathy
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/4
Other Adverse Events (participants affected / at risk) | 0/1 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No